CLINICAL TRIAL: NCT04532541
Title: Screening for Monogenic Lupus in Patients With Childhood Onset Systemic Lupus Erythematosus
Brief Title: Monogenic Lupus in Childhood Onset Systemic Lupus Erythematosus
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: Sunli-1
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Monogenic Lupus; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA anticoagulated peripheral blood is obtained from patients with childhood onset SLE and their biological parents. Samples are performed after parents' information and consent.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with childhood onset SLE: Participants in this group were derived from patients diagnosed with SLE at an age of less than 18 years old, and these patients were hospitalized in our center. Peripheral blood was collected from the patient and their biological parents for gene analysis to obtain the overall incidence of monogenic lupus in the cohort.
  Interventions: Other: Monogenic lupus screening

INTERVENTIONS:
Other: Monogenic lupus screening — This is an observational study, and there is no intervention. This study intends to obtain the incidence of monogenic lupus in childhood onset SLE through gene test and bioinformatic analysis.

SUMMARY:
The purpose of this study is to unravel the proportion of monogenic lupus in children onset Systemic lupus erythematosus (SLE), and to find out the diagnostic strategy for early detection of monogenic lupus.

DETAILED DESCRIPTION:
Childhood Systemic Lupus Erythematosus (SLE) is a common autoimmune disease in children, with a high incidence in Asia. Compared with adult SLE, childhood SLE is more likely to involve multiple systems, the treatment is more difficult, and mortality is relatively high. With the improvement of diagnosis and treatment of SLE, the prognosis of children with SLE continues to improve, but there are still a small number of patients who are ineffective to existing treatments. The pathogenesis of SLE is complicated, and more and more evidences confirm that genetic factors are involved in the pathogenesis of SLE. In recent years, the concept of "Monogenic Lupus" has been proposed internationally, and more than 30 single gene variants have been found to be related to the onset of SLE. Such patients are clinically in line with typical SLE or lupus-like syndrome, with common characteristics of a very young age of onset (mostly in infants and young children), and/or a family history of rheumatic immune diseases. It is a huge difficulty to early identify these patients at present, and it has not been generally accepted in the field of rheumatology in China.

In this research, about 200 patients with childhood onset SLE that meet the criteria for inclusion and exclusion were tested for gene analysis, and clinical data were collected and entered into the SLE cohort database. The incidence of monogenic lupus in childhood onset SLE will be unraveled. Based on clinical key words, such as early onset, male, family history of rheumatic diseases, blood system involvement, kidney involvement, the incidence of monogenic lupus in these single or multiple keyword combination will be calculated and compared to obtain an early, cost-effective diagnosis strategy for monogenic lupus.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet the following criteria will be allowed to participate in the study:

1. onset age: birth to 18 years;
2. meet the diagnostic criteria of SLE according to ACR(1997), or SLICC(2012), or EULAR/ACR (2019);
3. obtain parental consent.

Exclusion Criteria:

1. Lack of clinical data;
2. Unable to finish the follow-up.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants in this group were derived from patients diagnosed with SLE at an age of less than 18 years old, and these patients were hospitalized in our center.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Monogenic lupus in childhood onset SLE | Gene test will be conducted at the time of enrollment.
  The concept of "Monogenic Lupus" has been proposed internationally, diagnosed by gene test among patients with typical SLE or lupus-like syndrome, and more than 30 single gene variants have been currently found to be related to the onset of SLE. This study intends to detect monogenic lupus in patients with childhood-onset SLE through gene test and bioinformatic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No